CLINICAL TRIAL: NCT03458585
Title: Radiation Exposure Awareness From Patients Undergoing Nuclear Medicine Diagnostic 99mTc-MDP Bone Scans and 18F-FDG PET/CT Scans
Brief Title: Radiation Exposure Awareness From Patients Undergoing Nuclear Medicine Diagnostic Scans
Acronym: REA
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Royal Marsden NHS Foundation Trust (Other)
Collaborators: City, University of London (Other)
Responsible Party: Sponsor
Other Study IDs: CCR 4835
Record Dates: First submitted 2018-02-20; First posted 2018-03-08 (Actual); Last update posted 2018-06-29 (Actual); Status verified 2018-03

CONDITIONS: Skeletal Scintigraphy; FDG PET/CT
Keywords: ionising radiation; patient awareness; patient knowledge

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group 1: patients attending for a 99mTc-MDP bone scan.: Group 1: Patients will be approached after they had their injection for the bone scan procedure. Completion of questionnaire will take place during the three hour uptake period, before they have the scan.
  Interventions: Other: Self-administered questionnaire
- Group 2: patients attending for a 18F- FDG PET/CT scan.: Group 2: Patients will be approached and consented after they had their injection and scan for 18F- FDG PET/CT. Completion of questionnaire will take place immediately after patients have changed and wait to leave the department, while they wait for their scan to be checked .
  Interventions: Other: Self-administered questionnaire

INTERVENTIONS:
Other: Self-administered questionnaire — Self-administered questionnaire

SUMMARY:
This questionnaire is aimed at finding out if patients understand how much radiation they are being exposed to when they have a bone scan (99mTc-MDP)or an FDG PET/CT scan (18F-FDG PET/CT). This questionnaire is also interested in understanding if patients consider current leaflet information sent with appointment letter as sufficient to understand what the radiation dose from that scan is.

By collecting information on how much patients are aware and understand about radiation exposure, we can use this information to develop better guidance for medical staff who advise patients as well as clearer information leaflets for patients to assist in their understanding.

DETAILED DESCRIPTION:
Nuclear medicine uses ionizing radiation in order to diagnose and treat diseases and the different types of scans and therapies use different amounts and types of radiation which result in different exposures. For example in the UK the average natural background radiation levels is around 2.2 mSv and a Chest X-ray is about 0.014 mSv, which is equivalent to approximately 2.5 days of natural background radiation in the UK.

When undergoing clinical nuclear medicine scans such as 99mTC-MDP bone scans and 18F-FDG PET/CT scans, two of the most common procedures within nuclear medicine the current information made available to patients from clinicians and current information leaflets for both procedures may not be detailed enough to enable patients to understand about radiation exposure and make an informed decision to undergo the procedures.

With bone scans accounting for 27% of all conventional nuclear medicine procedures and 18F-FDG PET/CT scans accounting for 78% of total number of PET/CT procedures across the trust and similarly across the majority of nuclear medicine departments in England, this questionnaire aims to capture current knowledge and awareness of patients in terms of radiation exposure when they are referred for a nuclear medicine scan, their views on the current appropriateness of leaflets provided and how would they would prefer to receive that information.

This information will be used to potentially educate the medical staff on the need to correctly inform the patient with regards to radiation exposure; to standardize the information that is given to patients and to potentially design new information leaflets and request forms.

The current trust leaflets across all nuclear medicine procedures involving an injection of radiopharmaceutical have the same explanation under "Is there any risk from the radiation? The amount of radiation involved is small and similar to the amount used in some x-ray procedures." When in actual fact the exposure from a bone scan is around 4 mSv and the exposure from an 18F-FDG PET/CT is around 14 mSv which is significantly differently.

This is a cross sectional questionnaire study aimed at gaining a greater understanding of the patient perception and awareness of radiation exposure when undertaking a nuclear medicine 99mTc-MDP bone scan or 18F- FDG PET/CT scan.

Upon completion, patients will be given the fourth sheet of the cover letter with answers to questions on section 3. If patients have additional questions pertinent to the radiation exposure comparators they will be directed to the section on the cover letter where they can find more information regarding this subject. As appropriate questions will also be directed to the Principal Investigator who is Head of Radiation Protection at current Trust.

ELIGIBILITY:
Inclusion Criteria:

* Over the age of 18
* Group 1: undergoing a diagnostic bone scan within the Nuclear Medicine and PET/CT Department at The Royal Marsden Hospital
* Group 2: undergoing a diagnostic 18F- FDG PET/CT within the Nuclear Medicine and PET/CT Department at The Royal Marsden Hospital.

Exclusion Criteria:

* Previous participation in one group; (participants can only take part in one of the group questionnaires once).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Group 1: patients attending 99mTc-MDP bone scans. Group 2: patients attending 18F- FDG PET/CT scans.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2018-02-26 (Actual); Primary Completion 2018-12-31 (Estimated); Study Completion 2018-12-31 (Estimated)

PRIMARY OUTCOMES:
Self-reported knowledge of patients undergoing bone scan or FDG PET/CT | 9 months
  Self-administered questionnaire will be used to collect information on patient knowledge regarding exposure to ionising radiation when having the nuclear medicine scans such as bone scan or FDG PET/CT

SECONDARY OUTCOMES:
Qualitative assessment on current leaflets for bone scans and FDG PET/CT scans | 9 months
  Two open questions will be used to collect patients views and suggestions on information regarding doses of radiation used in the 2 procedures. Thematic analysis will be used to analyse data.
Demographic correlations with self-reported knowledge | 9 months
  Statistical correlations with age, gender, previous scans, level of education, confidence in completing medical forms and self-reported knowledge.

CONTACTS AND LOCATIONS:
Locations (1):
- The Royal Marsden Hospital NHS Trust Foundation, Sutton, Surrey, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided
Presentations and publications require authorisation by the CI who is responsible for the study.
  The International Committee of Medical Journal Editors (ICMJE) requires clinical trials to be entered onto a recognised registry before recruitment of the first patient, in order for the trial to be published in an ICMJE journal. This study will be registered on www.clinicaltrials.gov.
  A summary of the study findings will be available in the trust website.